# Investigating Participation Behavior: An Observational Study in Mild Cognitive Impairment Clinical Trials

An Informed Consent Form For Power Clinical Trial's Mild Cognitive Impairment Observational Study

Date: January 5, 2024

Introduction to the Informed Consent Form: A Brief Overview

This summary aims to provide an outline of our observational clinical study, highlighting its procedures, potential risks, and benefits for participants. While your consent is required, your participation is entirely voluntary, affording you the freedom to withdraw without any repercussions.

Our study aims to understand why patients with mild cognitive impairment choose to enroll, continue, or discontinue participation in clinical trials. The primary procedures include completing questionnaires and follow-up calls, tailored to minimize potential risks for participants.

Although direct medical benefits may not be immediate in this observational study, the gathered data will aid in identifying ways to enhance clinical trial participation rates, ultimately benefiting individuals affected by mild cognitive impairment.

The study's conclusions will provide crucial insights into the factors influencing clinical trial participation rates. Our objective is to refine recruitment strategies and bolster patient involvement in trials, leading to improved treatment options and outcomes for mild cognitive impairment sufferers. However, engaging in this study is voluntary, and declining participation will not impact your rights.

Thoroughly reviewing the consent form and seeking clarification on any concerns before making a decision is vital. Engaging in discussions with family, friends, advisors, and healthcare professionals is recommended to ensure an informed choice.

Participation remains entirely voluntary, with the right to withdraw at any time without facing consequences.

Factors Influencing Participation in Mild Cognitive Impairment Clinical Trials

Clinical trials are pivotal in advancing mild cognitive impairment treatments, yet concerns persist about participant representation. This study aims to probe into the determinants that sway patient decisions regarding participation, withdrawal, or re-engagement in mild cognitive impairment clinical trials. Uncovering these factors is crucial to enhance the relevance and efficacy of future research endeavors.

To ensure a comprehensive approach, our emphasis is on recruiting a diverse demographic pool. We aim to understand how variables like age, race, income, and education impact decision-making about participation. This gathered data aims to devise more effective approaches to engage underrepresented groups in forthcoming clinical trials.

Participation in this study is entirely voluntary, enabling individuals to withdraw without consequences. The study's procedures, involving questionnaire completion and follow-up calls, pose minimal risks. Prospective participants are strongly encouraged to thoroughly review the consent form and seek clarification for any queries.

Ultimately, this trial seeks to deepen our comprehension of the factors influencing mild cognitive impairment clinical trial participation. Heightening participation rates could accelerate the development of innovative treatments for this challenging ailment.

Exploring Mild Cognitive Impairment Patients' Participation in Clinical Trials

Through our observational clinical research, we aim to comprehend the factors influencing mild cognitive impairment patients' decisions regarding clinical trial participation—such as enrollment, withdrawal, and completion. We aim to involve potential participants from ongoing or concluded interventional trials, utilizing electronic medical records for identification purposes.

Upon expressing interest, our team will furnish a comprehensive consent form outlining the study's objectives and participant rights. Data collection involves regular biweekly questionnaires focusing on demographics, medical history, and the motives driving trial participation. Additionally, we plan to conduct comprehensive quarterly phone or video interviews to gain comprehensive participant insights.

The statistical analysis of the accumulated data aims to reveal the diverse factors shaping patient participation in clinical trials. Sharing our findings through conferences and academic publications aims to benefit all stakeholders involved in clinical trials.

We aim to leverage these insights to improve the design of future clinical studies for mild cognitive impairment patients, enhancing recruitment strategies and ensuring better retention rates.

Participation in this study is entirely voluntary, allowing individuals to withdraw without facing any consequences. Minimal risks involve the completion of questionnaires and follow-up interviews. Our readily accessible research team can promptly address any queries or concerns.

Evaluating Potential Risks in Mild Cognitive Impairment Observational Studies

Participation in mild cognitive impairment observational studies doesn't involve experimental treatments, yet it might entail certain risks. These risks could involve breaches of privacy, emotional distress due to the study's subject matter, and potential negative consequences from trial-related procedures.

Before deciding to participate, it's essential to carefully review and comprehend the informed consent form and communicate any concerns with the research team. The team will provide comprehensive information regarding potential risks, the study's benefits, and safety measures implemented for the participants' protection.

Understanding the Potential Gains from Mild Cognitive Impairment Observational Trials

Participation in observational clinical trials focusing on mild cognitive impairment presents patients with a chance to contribute to medical progress and potentially

enhance future treatment alternatives. Even in the absence of experimental therapies, patients can receive comprehensive care throughout the study.

Before deciding to participate in the trial, patients should thoroughly assess potential benefits and risks, taking into consideration their individual circumstances and objectives. Seeking advice from healthcare providers and the research team is essential in making a well-considered decision.

### Key Considerations Influencing Your Participation Conclusion

Understanding that your involvement in a clinical trial could cease without your explicit consent is significant. Researchers or sponsors might conclude the trial due to various reasons, including study suspension, funding discontinuation, or if it's deemed beneficial for your well-being.

Moreover, your participation may end due to declining health, pregnancy, opting out following important updates, or failure to adhere to study guidelines. Considering these factors thoughtfully before deciding to participate in a clinical trial is highly important.

## Comparative Analysis of Mild Cognitive Impairment Trials

Engagement in mild cognitive impairment clinical trials is completely optional, affording participants the freedom to withdraw without encountering adverse consequences.

For a holistic perspective on <u>mild cognitive impairment research</u> globally, clinicaltrials.gov, managed by the National Institutes of Health (NIH), serves as an expansive repository of trials. Users can tailor their search based on location and specific medical conditions.

Moreover, Power's reference page offers an updated compilation of active <u>mild cognitive</u> <u>impairment clinical trials</u> presently seeking participants.

# Exploring Clinical Trial Diversity Through Online Sources

Various online platforms cater to individuals seeking in-depth knowledge about clinical trial diversity. Here are a couple of articles that might attract your attention:

Woods-Burnham, Leanne, Jabril R. Johnson, Stanley E. Hooker, Fornati W. Bedell, Tanya B. Dorff, and Rick A. Kittles. "The role of diverse populations in US clinical trials." Med 2, no. 1 (2021): 21-24.

Masters, Joanna C., Jack A. Cook, Ginger Anderson, Gianluca Nucci, Anna Colzi, Marie-Pierre Hellio, and Brian Corrigan. "Ensuring diversity in clinical trials: The role of clinical pharmacology." Contemporary Clinical Trials 118 (2022): 106807.

These resources offer valuable insights into the challenges associated with clinical trial diversity and potential strategies to promote inclusivity within research studies.

### **Ensuring Confidentiality in Research Studies**

Maintaining the confidentiality of the data collected for this research is our paramount commitment. Although complete confidentiality cannot be universally guaranteed, robust measures have been implemented to safeguard it. Please note that legal obligations might necessitate the disclosure of personal information. Nonetheless, any research publications or presentations will prioritize your anonymity by refraining from disclosing your name or any personally identifying information.

Various entities, such as accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for purposes related to research, quality assurance, and data analysis.

In rare cases, we might require an "Authorization Form" detailing the use and sharing of your information for this study. Before sharing your information or research samples with Power researchers, other university institutions, or external commercial entities for future research, explicit consent will be obtained. Your confidential data will be handled securely and deleted as appropriate.

# Agreement to Informed Consent Terms

By providing your signature on this consent agreement, you acknowledge and accept the following terms:

- Thoroughly reading and comprehending this informed consent form, with encouragement to seek alternative viewpoints before making a decision.
- Satisfactory resolution of all your queries regarding the research project and its methodologies, ensuring you possess the necessary information for study participation.
- Contemplation of potential benefits, drawbacks, and alternatives associated with participation in the research.
- Assurance that your voluntary involvement in the research study will not hinder your legal rights.
- Timely communication of any significant updates that might impact your decision to continue participating in the research study.
- Receipt of this consent form allows you to address any remaining inquiries.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Researcher's Confirmation | | |
| In my role as the researcher, I have ensured the patient's queries were adequately attended to, facilitating a comprehensive grasp of the study. Additionally, I have reaffirmed that the patient's participation is voluntary and based on informed consent. | | |
| Signature of Researcher Who Received Consent | | |
| Name of Investigator | Signature of Investigator | Date |